CLINICAL TRIAL: NCT07067281
Title: A Comparative Study Between TAPP And Lichtenstein Techniques for Inguinal Hernia Surgery, A Prospective Study
Brief Title: A Comparative Study Between TAPP and Lichtenstein Techniques for Inguinal Hernia Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GSVM Medical College (Other)
Responsible Party: Principal Investigator, Shubham Chaubey, Junior Resident, Department of General Surgery, GSVM Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/BMHR/2024/34
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hernia Inguinal
Keywords: Trans abdominal preperitoneal repair; Operative time; Surgical site infection; Recurrence; Seroma; Mesh infection
MeSH Terms: conditions — Hernia, Inguinal; Surgical Wound Infection; Recurrence; Seroma | interventions — tetra-4-amidinophenoxypropane; Wound Healing

STUDY DESIGN:
Intervention Model Description: Randomized parallel Group,Active trial with computer generated randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lichtenstein Techniques for Inguinal Hernia surgery using as conventional method (Active Comparator): Participants randomized to this arm will undergo open Lichtenstein tension-free mesh repair for inguinal hernia under regional (spinal) or local anesthesia. A standard polypropylene mesh will be placed over the inguinal canal posterior wall and fixed to the inguinal ligament and conjoint tendon using non-absorbable sutures. The procedure is performed through a single inguinal incision. Patients will receive perioperative analgesia and standard postoperative care. This technique serves as the control group, reflecting conventional open hernia repair.
  Interventions: Procedure: Lichtenstein Tension-Free Mesh Hernioplasty
- TAPP Repair (Experimental): Participants in this arm will undergo laparoscopic Transabdominal Preperitoneal (TAPP) repair of inguinal hernia under general anesthesia. A standard 3-port laparoscopic technique will be used. After accessing the preperitoneal space, a large polypropylene mesh will be placed to cover the myopectineal orifice and fixed using tacks or glue. The peritoneal flap will be closed using absorbable sutures or staplers. Patients will receive standard laparoscopic postoperative care. This arm represents the minimally invasive surgical option.
  Interventions: Procedure: Laparoscopic Transabdominal Preperitoneal (TAPP) Repair

INTERVENTIONS:
Procedure: Lichtenstein Tension-Free Mesh Hernioplasty — Open surgical repair of inguinal hernia using a tension-free mesh technique. A standard polypropylene mesh is placed over the posterior wall of the inguinal canal and fixed with non-absorbable sutures under spinal or local anesthesia. This is a conventional method widely used in open hernia surgery.
  Arms: Lichtenstein Techniques for Inguinal Hernia surgery using as conventional method
Procedure: Laparoscopic Transabdominal Preperitoneal (TAPP) Repair — Laparoscopic approach to inguinal hernia repair performed under general anesthesia. Three ports are used to access the abdominal cavity, and a peritoneal flap is created to place a large polypropylene mesh in the preperitoneal space. The mesh is fixed with tacks or glue, and the peritoneal flap is closed. This minimally invasive method is designed to reduce postoperative pain and enhance recovery.
  Arms: TAPP Repair

SUMMARY:
This study is comperative study between TAPP And Lichtenstein Techniques for Inguinal Hernia surgery.The Lichtenstein tension-free open hernioplasty involves placing a tailored polypropylene mesh over the inguinal canal defect, secured to ligament and oblique fascia under local/regional anesthesia.Transabdominal Preperitoneal (TAPP) hernia repair uses laparoscopic access via three ports (umbilicus and bilateral midclavicular lines), incises and closes a peritoneal flap, and places a large mesh in the preperitoneal space. Compression between these two procedure in terms of intraoperative ,postoperative complications and Long term follow up for recurrence of Hernia.

DETAILED DESCRIPTION:
Comperative study between TAPP And Lichtenstein Techniques for Inguinal Hernia surgery.

Worldwide, inguinal hernia repair is one of the commonest surgeries. The best treatment option to primary hernia has been investigated, but there still remains lack of evidence about the ideal approach.

Therefore, this study aimed to compare the outcomes of inguinal hernia repair using Trans abdominal Pre peritoneal procedure(TAPP) & Lichtenstein techniques. Primary outcomes are Operative time , Surgical site infection , Seroma , post operative ileus , bowel injury ,mesh infection , recurrence and quality of life .

ELIGIBILITY:
Inclusion Criteria: 1. 5 -80 years 2. Any gender 3. Direct Hernia 4. Indirect hernia

-

Exclusion Criteria: 1 . Patient who are not fit for general anesthesia 2. Patient with lateral hernia 3 . Patient with complicated inguinal hernia like instructed and strangulated hernia

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Operative time | Intraoperative (measure during surgical procedure on day1)
  Total duration of surgery in minutes, measure skin incision to reversal of pneumoperitoneum

SECONDARY OUTCOMES:
Postoperative ileus | Up to 5 days
  Delayed return of bowel function by flatus or bowel movement, abdominal distention or need for nasogastic tube decompression
Surgical site infection | Up to 30 days post operation
  Superficial and deep wound infection including erythema , discharge or wound dehiscence
Hospital stay | From date of surgery untill discharge , assessed upto 14days
  Total number of days the date of operation to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Shubham Chaubey, Principle investigator, MBBS, Principal Investigator — GSVM MEDICAL COLLEGE KANPUR
Locations (1):
- Ganesh Shankar vidhyapthi Memorial Medical college kanpur, Kanpur, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participants( IPD ) related to operative time, hospital stay and post operative complications
Supporting Information: CSR
Time Frame: 6 months after publication of results for 2 years
Access Criteria: Qualifed researchers upon reasonable request